CLINICAL TRIAL: NCT04968327
Title: Effect of Micro-osteoperforations on the Rate of Canine Retraction; A Split-mouth Randomized Controlled Clinical Trial
Brief Title: Micro-osteoperforations on the Rate of Canine Retraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Canine retraction2020
Record Dates: First submitted 2021-07-05; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Intervention Model Description: split-mouth
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micro-osteoperforations (Experimental)
  Interventions: Other: Micro-osteoperforations (MOPs); Other: Conventional canine retraction
- Canine retraction (Active Comparator)
  Interventions: Other: Conventional canine retraction

INTERVENTIONS:
Other: Micro-osteoperforations (MOPs) — MOPs included shallow perforations of the buccal cortical plate surrounding the tooth that requires orthodontic tooth movement, with no flap reflection was performed using a surgical bur using the special calibrated device called PROPEL
  Arms: Micro-osteoperforations
Other: Conventional canine retraction — using nickel-titanium (NiTi) closed coil-springs delivering a force of 150 grams per side

SUMMARY:
the study aimed to clinically evaluate the effect of micro-osteoperforations on the rate of tooth movement, as evaluated by its effect on the rate of canine retraction.

DETAILED DESCRIPTION:
Ten adult patients requiring maxillary first premolars' extraction were enrolled in this split-mouth randomized controlled clinical trial.

Micro-osteoperforations were randomly assigned to one side of the maxillary arch at the canine-premolar region, and the contralateral side served as the control.

Mini-screws were used for anchorage reinforcement, and canine retraction was performed using nickel-titanium closed coil springs, delivering a force of 150 grams per side.

The primary outcome was the measurement of canine retraction rate throughout the study period from digital dental models obtained every 3 weeks.

The secondary outcome was the detection of possible canine tipping during retraction.

ELIGIBILITY:
Inclusion Criteria:

* healthy systemic condition with no chronic diseases
* no previous orthodontic treatment
* adequate oral hygiene
* have a healthy periodontium
* signed an informed consent

Exclusion Criteria:

* have a chronic disease
* previous orthodontic treatment
* poor oral hygiene or periodontal conidition

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Rate of canine retraction | 12 weeks
  measurements were recorded from digital dental models every 3 weeks

SECONDARY OUTCOMES:
Measurment of canine tipping | 12 weeks
  Tipping of the maxillary canine during retraction was also evaluated from digital dental models

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt